CLINICAL TRIAL: NCT07274098
Title: A Randomised Controlled Pilot Study of the Effectiveness of a VR Headset on Post Operative Relaxation, Anxiety and Pain in Patients Undergoing Elective Laparoscopic Colorectal Surgery
Brief Title: To Test Effectiveness of Virtual Reality on Post Operative Patients 'VR-RAP@
Acronym: VR-RAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: East Kent Hospitals University NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 338543
Record Dates: First submitted 2025-11-26; First posted 2025-12-10 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-11

CONDITIONS: Colo-rectal Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (No Intervention): This arm received Standard care
- Virtual Reality (Experimental): This arm receives the VR intervention Virtual Reality
  Interventions: Device: Virtual reality

INTERVENTIONS:
Device: Virtual reality — If randomised to VR then the patient will wear the unit twice a day, morning and afternoon, if possible, before the ward drug round, for a maximum of 5 days whilst they are in hospital. The number of days will depend on the length of time the participant is in hospital post surgery.
  Arms: Virtual Reality

SUMMARY:
Virtual reality (VR) headsets (like those used in gaming) allow users to feel immersed in an artificial 3 dimensional environment. The user is able to look around within the environment and interact with it.

Virtual reality has been used extensively in video games and also in training eg in flight simulators used to train pilots.

There is now a growing use of VR in a clinical setting as virtual reality environments have been designed to help users relax and reduce anxiety or distract and reduce pain. Trials have shown that these can work in many situations including helping relax staff who are working in highly stressful situations, or to distract and help reduce pain in patients following injuries or during minor operations. The relaxation environments use pictures and sounds to create calm environments and can guide users in breathing exercises which help calm and relax. This study is to investigate whether it will be possible to do a study using a VR headset with a relaxation experience, in the days following abdominal surgery that leads to a reduction in anxiety and pain.

Two groups of patients will be studied, one group will use the head set twice a day for up to 5 days and the other will not. They will record their pain and anxiety on a scale of 1 to 10 every day. The amount of pain reducing medicines that they need will also be recorded. The patients will be randomly divided into the 2 groups, they will not get to choose.

The researchers will see whether patients are happy to use the headsets following surgery and at the end of the study, the pain and anxiety scores for the group which used the VR headset will be compared with the scores for the group that didn't.

DETAILED DESCRIPTION:
Potential participants will be identified within the Multi Disciplinary Team (MDT) meetings and review of theatre lists by the Chief Investigator or the relevant delegated research staff. They will be approached before surgery by a member of the research team (who are part of the clinical care team) when they have their pre-assessment appointment or contacted when they have been deemed eligible .

If they are interested in being involved in the study they will be given a copy of the Participant information sheet (PIS) and given the opportunity to ask any initial questions. Patients will have ample time and opportunity to review and consider the PIS In the days prior to surgery they will be contacted to see if they would like to take part and ask any questions.

If they do want to take part, they will give consent to a member of the research study team any time before surgery.

Once consented, the participants will be shown how to use the equipment and the relaxation courses that are available . This will take place in hospital either at an appointment or on day of surgery The participant will be randomised on the day of surgery to either standard of care (SOC) or VR. Randomisation will not take place before the day of surgery in case the surgery is cancelled or doesn't go ahead for other reasons.

On the day of surgery, before surgery, all participants will complete a questionnaire, , about their mood, anxiety levels and pain score using visual analogue scales (VAS). This will be the baseline data.

Data will be collected on the day of surgery post surgery and from day 1 after surgery. Ideally this will be before the ward drug round. This will ensure that the effect on pain levels of using VR can be fairly measured. Data will be collected on Pain score, Anxiety levels, medication required. If randomised to VR then the patient will wear the unit twice a day, morning and afternoon, if possible, before the ward drug round, for a maximum of 5 days whilst they are in hospital. The number of days will depend on the length of time the participant is in hospital post surgery. All participants will complete a questionnaire where they will also be asked about their mood, anxiety levels and pain score using visual analogue scales (VAS) twice a day, morning and afternoon, until discharge or for a maximum of 5 days whilst they are in hospital. Those randomised to the VR arm will also be asked which scenario they watched, for how long and how comfortable they found the headset On day 14 (+/- 1)after surgery, when most participants should have returned home, they will be contacted and asked to complete the questionnaires for a final time.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 years and above Having elective laparoscopic colorectal surgery Patients who are able to understand English and can understand the Participant Information Sheet and give informed consent to take part in the study.

Exclusion Criteria:

presence of motion sickness

* stroke
* Severe nausea
* isolation status for infection control
* neurological conditions i.e. dementia, seizure, epilepsy
* Suffering from delirium or acute confusional state
* Skin on face or head is broken i.e. head wounds or dermatological conditions
* Conversion to open surgery, if decided prior to consent
* Patients with severe visual impairment (i.e., not able to clearly see without glasses; patients with contact lenses will not be excluded).
* Inclusion in another trial to evaluate new ways of treating pain
* Use of strong opioids (i.e., morphine)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2025-04-16 (Actual); Primary Completion 2025-06-09 (Actual); Study Completion 2025-08-08 (Actual)

PRIMARY OUTCOMES:
Percent of participants in the virtual reality group who complete 80% of potential sessions (i.e. twice per day until discharge; maximum 5 days) | (i.e. twice per day until discharge; maximum 5 days)
  Percent of participants in the virtual reality group who complete 80% of potential sessions (i.e. twice per day until discharge; maximum 5 days)

CONTACTS AND LOCATIONS:
Locations (1):
- Kent and Canterbury Hospital, Canterbury, Kent, United Kingdom

IPD SHARING:
Plan to Share IPD: No